CLINICAL TRIAL: NCT02447198
Title: Cannabidiol (CBD) and Pediatric Epilepsy
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0216; UL1TR001082 (NIH)
Record Dates: First submitted 2015-05-07; First posted 2015-05-18 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn up to 6 times. It will be centrifuged to collect the plasma. The plasma will be used to obtain concentration of cannabinols and anticonvulsant medications in order to perform pharmacokinetic calculations.
  All urine output for the first 8 hours after initial CBD dose will be collected.
Oversight: Data Monitoring Committee: No

SUMMARY:
Legislation to allow medical marijuana has had a significant impact on the pediatric population of Colorado. There have been many reported different effects and properties of each of the over 60 known cannabinoids found in marijuana. The main exposures in pediatrics have involved the use of Cannabidiol (CBD) high- and Tetrahydrocannibinol (THC) low-content hash oil in children with epilepsy. The reported benefit of this oil is to have the anticonvulsant properties of CBD without the psychoactive components of THC. Human studies on the efficacy of CBD on epilepsy are few and limited.

The investigators' specific aims are the following:

* Specific Aim 1: Describe the plasma pharmacokinetics of Cannabidiol (CBD), Tetrahydrocannibinol (THC), and their respective metabolites in pediatric patients with epilepsy.
* Specific Aim 2: Describe the plasma pharmacokinetics of other antiepileptic drugs (AEDs) taken in conjunction with CBD in order to evaluate drug interactions.
* Specific Aim 3: Describe parental perception of efficacy of CBD on control of epilepsy.

The investigators will recruit children and their parents who are currently using or plan to use CBD for their seizure disorder. This study will NOT be providing patients with CBD. Consenting subjects will undergo a number of blood and urine collection that will be analyzed to describe the pharmacokinetics and possible drug interactions of CBD in pediatric epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 1 month and < 18 years of age who use, or plan to use, orally administered CBD rich hash oil for treatment of epilepsy
* Parent/legal guardian accompanying patient who is >= 18 year of age and non-incarcerated.

Exclusion Criteria:

* Patients without epilepsy/seizure disorder as diagnosed by a neurologist
* Have known abnormalities in liver (AST, ALT, INR above normal range), or kidney function (creatinine above normal range)
* Patient is known to be pregnant at time of enrollment (however, guardians who may be pregnant can be included for survey completion)
* Patient is ward of the state
* Unable to provide verification of hash oil potency and content

Ages: 31 Days to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will recruit children and their parents who are currently using or plan to use CBD for their seizure disorder.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Describe the plasma pharmacokinetics of Cannabidiol (CBD), other antiepileptic drugs, Tetrahydrocannibinol (THC), and their respective metabolites in pediatric patients with epilepsy. | Change from baseline to 12 hours post CBD administration
  Blood samples will be obtained at 6 time periods: at baseline prior to the first dose of CBD and at the following time intervals after administration of CBD: 1 hour, 2 hour, 4 hour, 8 hour, and 12 hours after administration of CBD.
  Urine will be collected for first 8 hours to account for renal elimination of CBD and antiepileptics.

SECONDARY OUTCOMES:
Demographic Data | collected once at study visit
Medication History | collected once at study visit
CBD History | collected once at study visit
Describe parental perception of efficacy of CBD on control of epilepsy | collected once at study visit
  A parental survey will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: George Sam Wang, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Wang GS, Bourne DWA, Klawitter J, Sempio C, Chapman K, Knupp K, Wempe MF, Borgelt L, Christians U, Leonard J, Heard K, Bajaj L. Disposition of Oral Cannabidiol-Rich Cannabis Extracts in Children with Epilepsy. Clin Pharmacokinet. 2020 Aug;59(8):1005-1012. doi: 10.1007/s40262-020-00869-z. PMID 32048179